CLINICAL TRIAL: NCT00823316
Title: Phase 1/2 Study of Umbilical Cord Blood-Drived Mesenchymal Stem Cells Infusion for Promotion of Engraftment and Prevention of an Graft Rejection and Graft-versus-Host Disease After Unrelated Hematopoietic Stem Cell Transplantation.
Brief Title: Safety and Efficacy Study of Umbilical Cord Blood-Drived Mesenchymal Stem Cells to Promote Engraftment of Unrelated Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medipost Co Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP-CR-MSC003
Record Dates: First submitted 2009-01-13; First posted 2009-01-15 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-04

CONDITIONS: Acute Leukemia
Keywords: Mesenchymal Stem Cells; Allogeneic Transplantation; Engraftment; GvHD; Childhood; unrelated HSCT

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): at a dose of 1x1,000,000 hMSC/kg
  Interventions: Biological: Human umbilical cord blood-derived mesenchymal stem cells
- 2 (Experimental): at a dose of 5x1,000,000 hMSC/kg
  Interventions: Biological: Human umbilical cord blood-derived mesenchymal stem cells

INTERVENTIONS:
Biological: Human umbilical cord blood-derived mesenchymal stem cells — 1x1,000,000 hMSC/kg, IV after unrelated HSCT
  Other Names: PROMOSTEM
  Arms: 1
Biological: Human umbilical cord blood-derived mesenchymal stem cells — 5x1,000,000 hMSC/kg, IV after unrelated HSCT
  Other Names: PROMOSTEM
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of PROMOSTEM (human umbilical cord blood-derived mesenchymal stem cells) at a dose of 1 and 5x1,000,000 hMSC/kg in subject for the promotion of an engraftment and prevention of graft rejection and Graft-Versus-Host Disease after unrelated hematopoietic stem cell transplantation for children with acute leukemia.

DETAILED DESCRIPTION:
* Hematopoietic stem cell transplantation (HSCT) is a procedure in which progenitor cells capable of reconstituting normal bone marrow function are administered to a patient. This procedure has been used to treat adults and children with life-threatening hematological malignancies and congenital immunodeficiency disorders.
* In HSCT, therapeutic goal is an elimination of disease and enrichment of regenerating capacity to achieve engraftments resulting in continued generation of functional blood elements from the engrafted living cells. Transplantation of unrelated hematopoietic stem cells originating either from adult bone marrow or from peripheral blood often leads to graft-versus host-disease (GvHD), opportunistic infections and graft failure after transplantation.
* In HSCT, MSC have been used as a therapy for GvHD and other complications. The aim of MSC infusions in HSCT is to use the cells' immunomodulatory effects to promote engraftment and to reduce the immunological reactions giving rise to GvHD.
* There is a growing interest in co-transplantation of MSC and HSC to improve the donor outcome in the unrelated HSCT condition.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age 2~19 years old with plan to have unrelated hematopoietic stem cell transplantation with acute leukemia
2. Patient never has an experience of hematopoietic stem cell transplantation
3. Patient must have an acute leukemia with a complete remission.
4. Patients must have an ECOG 0~2.
5. No moderate or sever organ dysfunction : Ejection fraction > 45%; Creatinine <2.0 mg/ml; Serum bilirubin < 2 mg/ml; AST/ALT < 200 IU/L.
6. Patient must not have an transplantation with different source of hematopoietic stem cell such as bone marrow and cord blood.
7. Patient must not have an infection needed an administration of non-oral antibiotics.
8. No active severe infection derived form virus or fungus.
9. Each patient / patient's guardian must sign written informed consent.

Exclusion Criteria:

1. Patient has previously received hematopoietic stem cell transplantation.
2. Patient plans to have a related hematopoietic stem cell transplantation.
3. Patient has a severe internal disease.
4. Patient has enrolled another clinical trial study within last 4 weeks.

Ages: 2 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2008-08; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
- Day of neutrophil engraftment - Day of platelet engraftment - Evaluation of chimerism - Evaluation of engraftment rate | 28 and 100 days

SECONDARY OUTCOMES:
- AGVHD grade | 100 days

CONTACTS AND LOCATIONS:
Overall Officials: Hong Hoe Koo, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea